CLINICAL TRIAL: NCT03715426
Title: MKit: A Pilot Study Testing a Life Skills Application to Address Interpersonal Relationships in College
Brief Title: Testing a Life Skills Application to Address Interpersonal Relationships in College (MKit)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Michelle Munro-Kramer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00133004-A; KL2TR000434 (NIH); KL2TR002241 (NIH); 5R49CE002099-05 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2018-10-23 (Actual); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Sexual Violence; Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MKit WebApp Intervention (Experimental): The intervention arm will receive the usual standard of care training package for incoming students at the University of Michigan which includes: 1) Haven, an online module about healthy relationships and sexual violence completed before coming to campus; 2) Relationship Remix, an interactive peer-delivered program on healthy relationships and sexual violence; and 3) Change it Up, a bystander intervention educational theater performance delivered by student actors. In addition, they will receive access the MKit WebApp, which will give them access to content, goal setting, and resources for 14 topic areas.
  Interventions: Behavioral: MKit
- Standard of Care (No Intervention): The control arm will receive the usual standard of care training package for incoming students at the University of Michigan which includes: 1) Haven, an online module about healthy relationships and sexual violence completed before coming to campus; 2) Relationship Remix, an interactive peer-delivered program on healthy relationships and sexual violence; and 3) Change it Up, a bystander intervention educational theater performance delivered by student actors.

INTERVENTIONS:
Behavioral: MKit — MKit is a web-based application that uses a life-skills approach to address healthy relationships and sexual violence. It includes 14 tiles which incorporate information, goal setting, and resources.
  Arms: MKit WebApp Intervention

SUMMARY:
This study utilizes implementation science principles to culturally adapt a pre-existing web-based application (WebApp) for use with college students. The ADAPT-ITT process will be utilized to adapt the WebApp to a diverse (race, ethnicity, gender/sexual identity) college population with a focus on life skills and holistic self-care as reinforcement to currently available primary prevention programming available to incoming students. The study hypothesis is that the adapted WebApp will be usable, acceptable, and students will be willing to use it as a reinforcement to current university primary prevention programming. The study team will also monitor retention of participants over the academic year. This is a repeat pilot test to evaluate changes implemented to the WebApp after the initial pilot during the 2017-2018 academic year.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled as a student at the participating university (University of Michigan)
* Age 18 or older
* Willing to participate in the study
* Able to speak and read English
* Participated in Relationship Remix at the University of Michigan at residence halls during the Fall of 2018.
* Enroll with your University of Michigan email.

Exclusion Criteria:

* Did not complete the Relationship Remix session.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Munro-Kramer, PhD,CNM,FNP, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fincham FD, Cui M, Braithwaite S, Pasley K. Attitudes toward intimate partner violence in dating relationships. Psychol Assess. 2008 Sep;20(3):260-9. doi: 10.1037/1040-3590.20.3.260. PMID 18778162
- [Result] Heron SL, Thompson MP, Jackson E, Kaslow NJ. Do responses to an intimate partner violence screen predict scores on a comprehensive measure of intimate partner violence in low-income black women? Ann Emerg Med. 2003 Oct;42(4):483-91. doi: 10.1067/s0196-0644(03)00718-2. PMID 14520319
- [Result] Brook J. SUS - A quick and dirty usability scale. In P. W. Jordan, B. Thomas, B. A. Weerdmeester, McClelland (Eds.). Usability evaluation in industry. London: Taylor & Francis; 1996:189-194.
- [Result] Koss MP, Abbey A, Campbell R, Cook S, Norris J, Testa C, Ullman S, West C, White J. Revising the SES: A collaborative process to improve assessment of sexual aggression and victimization. Psychology Women Quarterly 31:357-370, 2007. doi:10.13072/midss.279
- [Result] Busch NB. Outcome measures for sexual assault services in Texas. The University of Texas at Austin; 2003. Retrieved from https://s3.us-east-2.amazonaws.com/wcasa/old-website-resources/Evaluation-Selecting%2BIndicators-Measure%2BDatabase%2B15.%2BOutcome_Measures_Texas%2BManual.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the mandatory primary prevention program, Relationship Remix, offered to all incoming students at the University of Michigan. We specifically recruited from October 21, 2018 - November 11, 2018 from Alice Lloyd Residence Hall (control) and Couzens and Fletcher Residence Halls (intervention).
Pre-assignment Details: In the MKit WebApp Intervention group, 1 potential participant did not complete the baseline survey. In the Standard of Care group, 4 potential participants did not complete the baseline survey. All of these potential participants were therefore not considered enrolled for the purposes of outcome analyses.
Period: Overall Study
Arm/Group | MKit WebApp Intervention | Standard of Care
Started | 133 | 117
1-Month Follow-Up Survey | 113 | 97
4-Month Follow-Up Survey | 112 | 92
Completed | 112 | 92
Not Completed | 21 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MKit WebApp Intervention | Standard of Care | Total
Number analyzed (Participants) | 133 | 117 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.19 (0.617) | 18.17 (0.460) | 18.18 (0.548)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 53 | 52 | 105
  Female | 75 | 64 | 139
  Trans Female/Trans Woman | 1 | 0 | 1
  Trans Male/Trans Man | 0 | 0 | 0
  Genderqueer/Gender Nonconforming | 1 | 0 | 1
  Different Identity | 2 | 0 | 2
  Prefer Not to Disclose | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 67 | 65 | 132
  Black/African American | 12 | 3 | 15
  Hispanic/Latino/Spanish | 5 | 7 | 12
  Middle Eastern/North African | 6 | 1 | 7
  Asian | 34 | 34 | 68
  Native Hawaiian/Other Pacific Islander | 1 | 0 | 1
  Multiple Ethnicities/Other | 8 | 7 | 15
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual or Straight | 114 | 103 | 217
  Gay or Lesbian | 3 | 3 | 6
  Bisexual | 7 | 8 | 15
  Something Else | 3 | 2 | 5
  Prefer not to disclose | 6 | 1 | 7
Year in School [Count of Participants; unit: Participants]
  Freshman | 123 | 111 | 234
  Sophomore | 6 | 4 | 10
  Junior | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Usability of the MKit WebApp as Assessed by the 10-item System Usability Scale
Description: Usability of the MKit WebApp will be measured using the 10-item System Usability Scale. Participants in the experimental group will complete the System Usability Scale, which is a 10 item questionnaire with responses that are rated from 1 (Strongly Disagree) to 5 (Strongly Agree) regarding use of the MKit WebApp. To get a final score: 1) First, one is subtracted from the score of the odd items; 2) Second, the responses are subtracted from 5 for the even-numbered items; 3) Then the responses are summed and multiplied by 2.5 to get a range of 0-100. A score above 68 is considered above average for perceived usability.
Time Frame: 1-month
Population: Only intervention participants were asked the items on the System Usability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 113
score on a scale | 64.36 (20.86)

2. Primary Outcome: Usability of the MKit WebApp as Assessed by the 10-item System Usability Scale
Description: as for outcome 1
Time Frame: 4-Months
Population: Only intervention participants were asked the items on the System Usability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 112
score on a scale | 62.08 (20.94)

3. Primary Outcome: Acceptability of the MKit WebApp as Assessed by the 5-item System Acceptability Scale
Description: The 5-item System Acceptability Scale (investigator created) will be used to evaluate the acceptability of the WebApp in the intervention group only. An investigator-created acceptability scale with 5-items will be used to measure acceptability. Four items are scored from 1 (Strongly Agree/Very Likely) to 5 (Strongly Disagree/Very Unlikely) and will be reverse coded. One item assesses the frequency of use of the WebApp from 1 (Never) to 5 (Multiple times a week). All five items will be summed for a total score. Scores range from 5-25, with higher scores indicating greater acceptability.
Time Frame: 1-Month
Population: Only intervention participants were asked the items on the System Acceptability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 113
score on a scale | 16.00 (2.91)

4. Primary Outcome: Acceptability of the MKit WebApp as Assessed by the 5-item System Acceptability Scale
Description: as for outcome 3
Time Frame: 4-Months
Population: Only intervention participants were asked the items on the System Acceptability Scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention
Number analyzed (Participants) | 112
score on a scale | 15.94 (3.32)

5. Secondary Outcome: 1-Month Retention
Description: The retention rate will be calculated based on how many participants in the intervention group have completed the follow-up surveys. A total retention rate (those retained/those enrolled) will be computed based on interaction with the WebApp.
Time Frame: 1-Month
Population: Retention was calculated based on the total number of participants that completed the Baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 133 | 117
Participants
  Completed 1-Month Survey | 113 | 97
  Did not complete 1-Month Survey | 20 | 20

6. Secondary Outcome: 4-Month Retention
Description: as for outcome 5
Time Frame: 4-Month
Population: Retention was calculated based on the total number of participants that completed the Baseline survey.
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 133 | 117
Participants
  Completed 4-Month Survey | 112 | 92
  Did not complete 4-Month Survey | 21 | 25

7. Other Pre Specified Outcome: 1-Month Sexual Victimization as Assessed by the 10-item Sexual Experiences Survey
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence victimization. The revised Sexual Experiences Survey - Short Form Victimization includes 10 items that are used to assess the frequency of seven victimization behaviors and then uses three questions to explore the sex of the perpetrator and if the participant believes they were raped. We will be items 1-7 to assess the number of times an individual has experienced victimization over the last 1 month from 0 to 3+ times. The results will be scored as a percentage of participants who have experienced each individual behavior and the percentage who report that they have experienced a rape.
Time Frame: 1-Month
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 113 | 97
Participants
  Victimization - Fondled, Kissed, or Rubbed Against: Experienced | 9 | 10
  Victimization - Fondled, Kissed, or Rubbed Against: Did not experience | 103 | 87
  Victimization - Fondled, Kissed, or Rubbed Against: Not Applicable | 0 | 0
  Victimization - Fondled, Kissed, or Rubbed Against: Missing | 1 | 0
  Victimization - Oral Sex: Experienced | 3 | 1
  Victimization - Oral Sex: Did not experience | 109 | 96
  Victimization - Oral Sex: Not Applicable | 0 | 0
  Victimization - Oral Sex: Missing | 1 | 0
  Victimization - Vaginal Sex: Experienced | 4 | 1
  Victimization - Vaginal Sex: Did not experience | 63 | 54
  Victimization - Vaginal Sex: Not Applicable | 45 | 41
  Victimization - Vaginal Sex: Missing | 1 | 1
  Victimization - Anal Sex: Experienced | 1 | 0
  Victimization - Anal Sex: Did not experience | 111 | 97
  Victimization - Anal Sex: Not Applicable | 0 | 0
  Victimization - Anal Sex: Missing | 1 | 0
  Victimization - Attempted Oral Sex: Experienced | 4 | 3
  Victimization - Attempted Oral Sex: Did not experience | 108 | 94
  Victimization - Attempted Oral Sex: Not Applicable | 0 | 0
  Victimization - Attempted Oral Sex: Missing | 1 | 0
  Victimization - Attempted Vaginal Sex: Experienced | 4 | 0
  Victimization - Attempted Vaginal Sex: Did not experience | 63 | 55
  Victimization - Attempted Vaginal Sex: Not Applicable | 45 | 41
  Victimization - Attempted Vaginal Sex: Missing | 1 | 1
  Victimization - Attempted Anal Sex: Experienced | 1 | 1
  Victimization - Attempted Anal Sex: Did not experience | 111 | 96
  Victimization - Attempted Anal Sex: Not Applicable | 0 | 0
  Victimization - Attempted Anal Sex: Missing | 1 | 0
  Victimization - Rape: Experienced | 6 | 1
  Victimization - Rape: Did not experience | 107 | 96
  Victimization - Rape: Not Applicable | 0 | 0
  Victimization - Rape: Missing | 0 | 0

8. Other Pre Specified Outcome: 4-Months Sexual Victimization as Assessed by the 10-item Sexual Experience Survey
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence victimization. The revised Sexual Experiences Survey - Short Form Victimization includes 10 items that are used to assess the frequency of seven victimization behaviors and then uses three questions to explore the sex of the perpetrator and if the participant believes they were raped. We will be items 1-7 to assess the number of times an individual has experienced victimization over the last 5 months from 0 to 3+ times. The results will be scored as a percentage of participants who have experienced each individual behavior and the percentage who report that they have experienced a rape.
Time Frame: 4-Months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
Participants
  Victimization - Fondled, Kissed, or Rubbed Against: Experienced | 7 | 9
  Victimization - Fondled, Kissed, or Rubbed Against: Did not experience | 104 | 83
  Victimization - Fondled, Kissed, or Rubbed Against: Not Applicable | 0 | 0
  Victimization - Fondled, Kissed, or Rubbed Against: Missing | 1 | 0
  Victimization - Oral Sex: Experienced | 4 | 2
  Victimization - Oral Sex: Did not experience | 107 | 90
  Victimization - Oral Sex: Not Applicable | 0 | 0
  Victimization - Oral Sex: Missing | 1 | 0
  Victimization - Vaginal Sex: Experienced | 1 | 3
  Victimization - Vaginal Sex: Did not experience | 67 | 49
  Victimization - Vaginal Sex: Not Applicable | 43 | 40
  Victimization - Vaginal Sex: Missing | 1 | 0
  Victimization - Anal Sex: Experienced | 1 | 0
  Victimization - Anal Sex: Did not experience | 110 | 92
  Victimization - Anal Sex: Not Applicable | 0 | 0
  Victimization - Anal Sex: Missing | 1 | 0
  Victimization - Attempted Oral Sex: Experienced | 3 | 1
  Victimization - Attempted Oral Sex: Did not experience | 108 | 91
  Victimization - Attempted Oral Sex: Not Applicable | 0 | 0
  Victimization - Attempted Oral Sex: Missing | 1 | 0
  Victimization - Attempted Vaginal Sex: Experienced | 0 | 1
  Victimization - Attempted Vaginal Sex: Did not experience | 67 | 51
  Victimization - Attempted Vaginal Sex: Not Applicable | 43 | 40
  Victimization - Attempted Vaginal Sex: Missing | 2 | 0
  Victimization - Attempted Anal Sex: Experienced | 0 | 0
  Victimization - Attempted Anal Sex: Did not experience | 111 | 92
  Victimization - Attempted Anal Sex: Not Applicable | 0 | 0
  Victimization - Attempted Anal Sex: Missing | 1 | 0
  Victimization - Rape: Experienced | 6 | 1
  Victimization - Rape: Did not experience | 105 | 91
  Victimization - Rape: Not Applicable | 0 | 0
  Victimization - Rape: Missing | 1 | 0

9. Other Pre Specified Outcome: 1-Month Sexual Violence Perpetration as Assessed by the 10-item Sexual Experience Survey
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence perpetration. The revised Sexual Experiences Survey - Short Form Perpetration includes seven items that are used to assess the frequency of perpetration of sexual violence behaviors and three questions that explore the sex of the victims and if the individual believes they have perpetrated a rape. We will be using these to assess the number of times an individual has perpetrated sexual violence over the last 1 month from 0 to 3+ times. The results will be scored as a percentage of participants who have perpetrated each individual behavior and the percentage who believe they have perpetrated a rape.
Time Frame: 1-Month
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 113 | 97
Participants
  Perpetration - Fondled, Kissed, or Rubbed Against: Perpetrated | 4 | 0
  Perpetration - Fondled, Kissed, or Rubbed Against: Did not perpetrate | 108 | 97
  Perpetration - Fondled, Kissed, or Rubbed Against: Missing | 1 | 0
  Perpetration - Oral Sex: Perpetrated | 1 | 0
  Perpetration - Oral Sex: Did not perpetrate | 111 | 97
  Perpetration - Oral Sex: Missing | 1 | 0
  Perpetration - Vaginal Sex: Perpetrated | 1 | 0
  Perpetration - Vaginal Sex: Did not perpetrate | 111 | 97
  Perpetration - Vaginal Sex: Missing | 1 | 0
  Perpetration - Anal Sex: Perpetrated | 1 | 0
  Perpetration - Anal Sex: Did not perpetrate | 111 | 97
  Perpetration - Anal Sex: Missing | 1 | 0
  Perpetration - Attempted Oral Sex: Perpetrated | 1 | 0
  Perpetration - Attempted Oral Sex: Did not perpetrate | 111 | 97
  Perpetration - Attempted Oral Sex: Missing | 1 | 0
  Perpetration - Attempted Vaginal Sex: Perpetrated | 1 | 0
  Perpetration - Attempted Vaginal Sex: Did not perpetrate | 111 | 97
  Perpetration - Attempted Vaginal Sex: Missing | 1 | 0
  Perpetration - Attempted Anal Sex: Perpetrated | 1 | 0
  Perpetration - Attempted Anal Sex: Did not perpetrate | 111 | 97
  Perpetration - Attempted Anal Sex: Missing | 1 | 0
  Perpetration - Rape: Perpetrated | 1 | 0
  Perpetration - Rape: Did not perpetrate | 112 | 97
  Perpetration - Rape: Missing | 0 | 0

10. Other Pre Specified Outcome: 4-Month Sexual Violence Perpetration as Assessed by the 10-item Sexual Experience Survey
Description: The 10-item Sexual Experiences Survey will be used to measure participants' experiences of sexual violence perpetration. The revised Sexual Experiences Survey - Short Form Perpetration includes seven items that are used to assess the frequency of perpetration of sexual violence behaviors and three questions that explore the sex of the victims and if the individual believes they have perpetrated a rape. We will be using these to assess the number of times an individual has perpetrated sexual violence over the last 4 months from 0 to 3+ times. The results will be scored as a percentage of participants who have perpetrated each individual behavior and the percentage who believe they have perpetrated a rape.
Time Frame: 4-Months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
Participants
  Perpetration - Fondled, Kissed, or Rubbed Against: Perpetrated | 2 | 1
  Perpetration - Fondled, Kissed, or Rubbed Against: Did not perpetrate | 109 | 91
  Perpetration - Fondled, Kissed, or Rubbed Against: Missing | 1 | 0
  Perpetration - Oral Sex: Perpetrated | 0 | 0
  Perpetration - Oral Sex: Did not perpetrate | 111 | 92
  Perpetration - Oral Sex: Missing | 1 | 0
  Perpetration - Vaginal Sex: Perpetrated | 0 | 0
  Perpetration - Vaginal Sex: Did not perpetrate | 111 | 92
  Perpetration - Vaginal Sex: Missing | 1 | 0
  Perpetration - Anal Sex: Perpetrated | 0 | 0
  Perpetration - Anal Sex: Did not perpetrate | 111 | 92
  Perpetration - Anal Sex: Missing | 1 | 0
  Perpetration - Attempted Oral Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Oral Sex: Did not perpetrate | 111 | 92
  Perpetration - Attempted Oral Sex: Missing | 1 | 0
  Perpetration - Attempted Vaginal Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Vaginal Sex: Did not perpetrate | 111 | 92
  Perpetration - Attempted Vaginal Sex: Missing | 1 | 0
  Perpetration - Attempted Anal Sex: Perpetrated | 0 | 0
  Perpetration - Attempted Anal Sex: Did not perpetrate | 111 | 92
  Perpetration - Attempted Anal Sex: Missing | 1 | 0
  Perpetration - Rape: Perpetrated | 1 | 0
  Perpetration - Rape: Did not perpetrate | 110 | 92
  Perpetration - Rape: Missing | 1 | 0

11. Other Pre Specified Outcome: 1-Month Sexual and Intimate Partner Violence Knowledge Questions Assessed With 20 Items Adapted From the Texas Education Program Participant Response Form
Description: Twenty knowledge questions about sexual and intimate partner violence adapted from the Texas Education Program Participant Response Form will be used to assess knowledge of healthy relationships, sexual violence, and intimate partner violence. The questions are scored from 1 (no knowledge) to 5 (a lot of knowledge) with higher scores indicating more knowledge. Possible sum scores range from 20 (no knowledge) to 100 (a lot of knowledge about all of the topics).
Time Frame: 1-Month
Population: Data for the 1-Month Knowledge scale were missing from 1 participant in the Intervention group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 97
score on a scale | 85.63 (12.09) | 82.77 (12.38)

12. Other Pre Specified Outcome: 4-Month Sexual and Intimate Partner Violence Knowledge Questions Assessed With 20 Items Adapted From the Texas Education Program Participant Response Form
Description: as for outcome 11
Time Frame: 4-Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
score on a scale | 84.05 (12.76) | 79.01 (14.09)

13. Other Pre Specified Outcome: Self-Efficacy of Protective Behaviors Related to Sexual and Intimate Partner Violence as Assessed by 15 Investigator Created Items
Description: Self-efficacy of protective behaviors related to sexual and intimate partner violence will be assessed using a questionnaire developed by the investigators. Participants will complete a 15 item questionnaire with responses ranging from 1 (not at all confident) to 7 (very confident) related to confidence in ability to handle situations related to sexual and intimate partner violence. The total score for each participant can range from 15 (not at all confident in any of the behaviors) to 105 (very confident in all behaviors).
Time Frame: 1-Month
Population: Data for the 1-Month Self-Efficacy scale were missing from 3 participants in the Intervention group and 5 participants in the Standard of Care group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 110 | 92
score on a scale | 93.45 (10.88) | 90.17 (11.50)

14. Other Pre Specified Outcome: Self-Efficacy of Protective Behaviors Related to Sexual and Intimate Partner Violence as Assessed by 15 Investigator Created Items
Description: as for outcome 13
Time Frame: 4-Months
Population: Data for the 4-Month Self-Efficacy scale were missing for 2 participants in the Intervention group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 110 | 92
score on a scale | 90.72 (13.07) | 88.33 (13.91)

15. Other Pre Specified Outcome: 1-Month Consensual Sexual Activity With 2 Investigator Created Items
Description: Two yes/no questions adopted from a colleague will be used to assess whether or not participants have ever engaged in sexual contact or intercourse that they found out was not consensual after the fact in the last 1 month. If they respond affirmatively then they will be asked an additional 14 descriptive questions about the event. Percent of students reporting ever engaging in sexual intercourse or contact that was not consensual will be reported.
Time Frame: 1-Month
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 113 | 97
Participants
  Non-Consensual Sexual Intercourse: Engaged in non-consensual sexual behavior | 2 | 1
  Non-Consensual Sexual Intercourse: Did not engage in non-consensual sexual behavior | 109 | 96
  Non-Consensual Sexual Intercourse: Missing | 2 | 0
  Non-Consensual Sexual Contact: Engaged in non-consensual sexual behavior | 2 | 2
  Non-Consensual Sexual Contact: Did not engage in non-consensual sexual behavior | 111 | 95
  Non-Consensual Sexual Contact: Missing | 0 | 0

16. Other Pre Specified Outcome: 4-Month Consensual Sexual Activity With 2 Investigator Created Items
Description: Two yes/no questions adopted from a colleague will be used to assess whether or not participants have ever engaged in sexual contact or intercourse that they found out was not consensual after the fact in the last 4 months. If they respond affirmatively then they will be asked an additional 14 descriptive questions about the event. Percent of students reporting ever engaging in sexual intercourse or contact that was not consensual will be reported.
Time Frame: 4-Months
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
Participants
  Non-Consensual Sexual Intercourse: Engaged in non-consensual sexual behavior | 2 | 2
  Non-Consensual Sexual Intercourse: Did not engage in non-consensual sexual behavior | 109 | 90
  Non-Consensual Sexual Intercourse: Missing | 1 | 0
  Non-Consensual Sexual Contact: Engaged in non-consensual sexual behavior | 1 | 1
  Non-Consensual Sexual Contact: Did not engage in non-consensual sexual behavior | 110 | 91
  Non-Consensual Sexual Contact: Missing | 1 | 0

17. Other Pre Specified Outcome: 1-Month Universal Violence Prevention Screening Protocol
Description: Thirteen yes/no questions from the Universal Violence Prevention Screening Protocol will be used to assess for personal experiences of intimate partner violence with the last 1 month. Each item will be evaluated individually and no total score will be computed.
Time Frame: 1-Month
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 113 | 97
Participants
  Been in a relationship in past 1 month: No | 74 | 71
  Been in a relationship in past 1 month: Yes | 39 | 26
  Been in a relationship in past 1 month: Not Asked | 0 | 0
  Been in a relationship in past 1 month: Missing | 0 | 0
  Slapped, kicked, pushed, choked, or punched: No | 37 | 23
  Slapped, kicked, pushed, choked, or punched: Yes | 1 | 3
  Slapped, kicked, pushed, choked, or punched: Not Asked | 74 | 71
  Slapped, kicked, pushed, choked, or punched: Missing | 1 | 0
  Forced or coerced you to have sex: No | 37 | 25
  Forced or coerced you to have sex: Yes | 1 | 1
  Forced or coerced you to have sex: Not Asked | 74 | 71
  Forced or coerced you to have sex: Missing | 1 | 0
  Threatened you with a weapon or blackmailed you: No | 38 | 25
  Threatened you with a weapon or blackmailed you: Yes | 0 | 1
  Threatened you with a weapon or blackmailed you: Not Asked | 74 | 71
  Threatened you with a weapon or blackmailed you: Missing | 1 | 0
  Made you afraid that you could be physically hurt: No | 38 | 25
  Made you afraid that you could be physically hurt: Yes | 0 | 1
  Made you afraid that you could be physically hurt: Not Asked | 74 | 71
  Made you afraid that you could be physically hurt: Missing | 1 | 0
  Repeatedly used words, yelled, or screamed at you: No | 37 | 25
  Repeatedly used words, yelled, or screamed at you: Yes | 1 | 1
  Repeatedly used words, yelled, or screamed at you: Not Asked | 74 | 71
  Repeatedly used words, yelled, or screamed at you: Missing | 1 | 0
  Controlled who/where you were allowed to see or go: No | 37 | 25
  Controlled who/where you were allowed to see or go: Yes | 1 | 1
  Controlled who/where you were allowed to see or go: Not Asked | 74 | 71
  Controlled who/where you were allowed to see or go: Missing | 1 | 0
  Minimized, denied, or normalized abusive behaviors: No | 38 | 25
  Minimized, denied, or normalized abusive behaviors: Yes | 0 | 1
  Minimized, denied, or normalized abusive behaviors: Not Asked | 74 | 71
  Minimized, denied, or normalized abusive behaviors: Missing | 1 | 0
  Threatened or abused important people or things: No | 38 | 25
  Threatened or abused important people or things: Yes | 0 | 1
  Threatened or abused important people or things: Not Asked | 74 | 71
  Threatened or abused important people or things: Missing | 1 | 0
  Used your identity to make you do something: No | 38 | 25
  Used your identity to make you do something: Yes | 0 | 1
  Used your identity to make you do something: Not Asked | 74 | 71
  Used your identity to make you do something: Missing | 1 | 0
  Used social media or texts to know where you are: No | 36 | 25
  Used social media or texts to know where you are: Yes | 2 | 1
  Used social media or texts to know where you are: Not Asked | 74 | 71
  Used social media or texts to know where you are: Missing | 1 | 0
  Monitored social media/required to share passwords: No | 37 | 25
  Monitored social media/required to share passwords: Yes | 1 | 1
  Monitored social media/required to share passwords: Not Asked | 74 | 71
  Monitored social media/required to share passwords: Missing | 1 | 0
  Sabotaged academic relationships/made feel unsmart: No | 38 | 25
  Sabotaged academic relationships/made feel unsmart: Yes | 0 | 1
  Sabotaged academic relationships/made feel unsmart: Not Asked | 74 | 71
  Sabotaged academic relationships/made feel unsmart: Missing | 1 | 0

18. Other Pre Specified Outcome: 4-Month Universal Violence Prevention Screening Protocol
Description: Thirteen yes/no questions from the Universal Violence Prevention Screening Protocol will be used to assess for personal experiences of intimate partner violence with the last 4 months. Each item will be evaluated individually and no total score will be computed.
Time Frame: 4-Month
Population: All of the "Not Asked" individuals (following the first question) were those who reported that they were not in a relationship in the past 4 months in the first question.
Measure: Count of Participants; unit: Participants
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
Participants
  Been in a relationship in past 4 months: No | 71 | 69
  Been in a relationship in past 4 months: Yes | 41 | 23
  Been in a relationship in past 4 months: Not Asked | 0 | 0
  Slapped, kicked, pushed, choked, or punched: No | 38 | 23
  Slapped, kicked, pushed, choked, or punched: Yes | 3 | 0
  Slapped, kicked, pushed, choked, or punched: Not Asked | 71 | 69
  Forced or coerced you to have sex: No | 37 | 23
  Forced or coerced you to have sex: Yes | 4 | 0
  Forced or coerced you to have sex: Not Asked | 71 | 69
  Threatened you with a weapon or blackmailed you: No | 41 | 23
  Threatened you with a weapon or blackmailed you: Yes | 0 | 0
  Threatened you with a weapon or blackmailed you: Not Asked | 71 | 69
  Made you afraid that you could be physically hurt: No | 41 | 23
  Made you afraid that you could be physically hurt: Yes | 0 | 0
  Made you afraid that you could be physically hurt: Not Asked | 71 | 69
  Repeatedly used words, yelled, or screamed at you: No | 39 | 23
  Repeatedly used words, yelled, or screamed at you: Yes | 2 | 0
  Repeatedly used words, yelled, or screamed at you: Not Asked | 71 | 69
  Controlled who/where you were allowed to see or go: No | 39 | 23
  Controlled who/where you were allowed to see or go: Yes | 2 | 0
  Controlled who/where you were allowed to see or go: Not Asked | 71 | 69
  Minimized, denied, or normalized abusive behaviors: No | 37 | 23
  Minimized, denied, or normalized abusive behaviors: Yes | 4 | 0
  Minimized, denied, or normalized abusive behaviors: Not Asked | 71 | 69
  Threatened or abused important people or things: No | 41 | 23
  Threatened or abused important people or things: Yes | 0 | 0
  Threatened or abused important people or things: Not Asked | 71 | 69
  Used your identity to make you do something: No | 40 | 23
  Used your identity to make you do something: Yes | 1 | 0
  Used your identity to make you do something: Not Asked | 71 | 69
  Used social media or texts to know where you are: No | 40 | 23
  Used social media or texts to know where you are: Yes | 1 | 0
  Used social media or texts to know where you are: Not Asked | 71 | 69
  Monitored social media/required to share passwords: No | 40 | 23
  Monitored social media/required to share passwords: Yes | 1 | 0
  Monitored social media/required to share passwords: Not Asked | 71 | 69
  Sabotaged academic relationships/made feel unsmart: No | 40 | 23
  Sabotaged academic relationships/made feel unsmart: Yes | 1 | 0
  Sabotaged academic relationships/made feel unsmart: Not Asked | 71 | 69

19. Other Pre Specified Outcome: 1-Month Intimate Partner Violence Attitude Scale
Description: Seventeen questions from the Intimate Partner Violence Attitude Scale - Revised will be used to assess for participant's attitudes related to intimate partner violence. Possible responses are on a Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree) with some items requiring reverse coding. Potential sum scores range from 17 to 85 with higher scores indicating a more favorable attitude towards intimate partner violence behaviors.
Time Frame: 1-Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 113 | 97
score on a scale | 26.80 (9.05) | 28.81 (9.72)

20. Other Pre Specified Outcome: 4-Month Intimate Partner Violence Attitude Scale
Description: as for outcome 19
Time Frame: 4-Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MKit WebApp Intervention | Standard of Care
Number analyzed (Participants) | 112 | 92
score on a scale | 27.70 (9.52) | 28.60 (10.43)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Since this was an anonymous study, adverse events were defined as those reported to study staff.
Arm/Group | MKit WebApp Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/133 | 0/117
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/117
Other Adverse Events (participants affected / at risk) | 0/133 | 0/117

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/26/NCT03715426/Prot_SAP_000.pdf